CLINICAL TRIAL: NCT06075472
Title: The Effect of Inspiratory Muscle Training on Balance and Postural Control in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tuğçe Duman Özkan, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MarmaraU_DumanOzkan_01
Record Dates: First submitted 2022-12-29; First posted 2023-10-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: balance; inspiratory muscle training; postural control
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): IMT: Inspiratory Muscle Training. Five days per week, 30 minutes per day.
  Interventions: Other: Inspiratory Muscle Training; Other: Balance Exercises
- Control Group (Active Comparator): Balance exercises: It has been specially designed for the patient.
  Interventions: Other: Balance Exercises

INTERVENTIONS:
Other: Inspiratory Muscle Training — Inspiratory muscle training (IMT) is a therapeutic technique which involves specific training of respiratory muscles to yield improvements in inspiratory muscle strength and respiratory function.
  Arms: Treatment Group
Other: Balance Exercises — Balance exercises involve functional movements at the individual's maximum level of independence.

SUMMARY:
The goal of this study is to investigate the effect of inspiratory muscle training (IMT) in Multiple Sclerosis (MS) patients on balance and postural control. The main question it aims to answer are:

• Is IMT effective in improving balance and postural control in MS patients? Participants will be randomly divided into two groups. One group will be given only balance exercises. The other group will be given IMT treatment in addition to balance exercises.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory, demyelinating and neurodegenerative disease of the central nervous system (CNS). MS is a disease that usually progresses with attacks and can lead to progressive disability and severely restrict the quality of life in patients due to the accumulation of sequelae after attacks or the development of a progressive degenerative process. Somatosensory findings, motor findings, postural control-balance and coordination disorders, bladder-intestinal problems, visual, cognitive and psychiatric findings, fatigue and sleep disorders are seen in patients related to the CNS involvement site.

Balance, one of the International Classification of Functioning headings, is a skill included in activity and participation, expressing the body's ability to maintain its upright position against gravity, and reflects stability limits. Balance impairment is one of the most common problems in patients with MS and is one of the factors that cause disability. Lesions in the brain stem and cerebellum cause loss of postural control and balance. There are many causes of loss of balance: visual symptoms, optic neuritis, vestibular changes, somatosensory changes, ventromedial tract lesion, tone changes, loss of muscle strength, incoordination.

Respiratory dysfunction in individuals with MS is an important problem that starts from the early period of the disease, increases in severity with the progression of the disability and causes mortality. Considering the pathophysiology of respiratory problems in MS, unlike other neuromuscular diseases, demyelinating lesions are found and spread in one or more areas related to breathing in the brain and spinal cord. The location and size of the plaques were associated with muscle weakness.

One of the methods used in the field of pulmonary rehabilitation in MS patients is Inspiratory Muscle Training (IMT). The muscles responsible for primary inspiration are the diaphragm, external intercostal muscles, and scalene muscles. Inspiratory muscle training increases inspiratory muscle strength, type 1 muscle fibers, reduces dyspnea, increases maximum minute ventilation and 6-minute walking distance and quality of life. It is usually applied at 30% of the maximal inspiratory pressure (MIP) value for 30 minutes a day.

The effect of the core muscles is great in providing balance and postural control. The diaphragm forms the roof of the core muscles and plays an important role in the mobility of the thorax. Training the diaphragm muscle, like other muscles, is important for maintaining dynamic and static balance. IMT can help stabilize thoracic mobility by strengthening the diaphragm and scalene muscles, contributing to the stability of chest movements and improving transfer skills.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of relapsing-remitting MS with an EDSS of 1.5-5.5
* Having a Mini Mental Test score greater than 24
* Being between the ages of 18-65

Exclusion Criteria:

* Having a neurological disease other than MS
* Having an attack while working
* Problems other than MS that may affect balance
* Have a diagnosis of cardiac or pulmonary disease that will affect breathing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Mini-BesTEST | Fifteen minutes
  Mini-BESTest consists of 14 items divided into four subsections. In the Mini-BESTest evaluation, each item receives a three-point score.
  rated on an ordinal scale (0= lowest function ranging from level to 2= Normal function level). The total score is the sum of the scores obtained from these items. and ranges from 0 (worst) to 28 (best).
Trunk Impact Scale | Ten minutes
  The Trunk Impact Scale (TIS) consists of three subscales: static sitting balance, dynamic sitting balance and co-ordination. Each subscale contains between three and ten items. The TIS score ranges from a minimum of 0 to a maximum of 23.

SECONDARY OUTCOMES:
Falls Efficacy Scale International | Fifteen Minutes
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the level of concern about falling during 16 social and physical activities inside and outside the home whether or not the person actually does the activity. The level of concern is measured on a four-point Likert scale (1=not at all concerned to 4=very concerned).
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Twenty minutes
  The Multiple Sclerosis Quality of Life-54 (MSQOL-54) was developed by using the RAND 36-item Health Survey 1.0 (SF-36) as a generic core measure, to enable comparisons of health-related quality of life (HRQOL) of patients with multiple sclerosis to those of other patient populations and to the general population.
  To enhance comparisons within groups of multiple sclerosis patients, these items were supplemented with 16 additional items in the areas of health distress, sexual function, satisfaction with sexual function, overall quality of life, cognitive function, energy, pain, and social function.
  The final measure, the MSQOL-54 Instrument, contains 54 items.
Activities-Specific Balance Confidence Scale | Ten Minutes
  The Activities-Specific Balance Confidence (ABC) Scale is a patient-reported outcome measure that asks individuals to rate how confident they are that they will not lose their balance while performing 16 different activities.
  The ABC Activities range from common tasks like walking around the house to less common and more challenging situations, like stepping off of a moving escalator while carrying packages. The patient is asked to rate their confidence in their balance, while performing 16 activities, on a percentage scale of 0 to 100, where 0 is a certainty of falling or becoming unstable and 100 is complete confidence in the patient's own ability to stay balanced.
Two minutes walking test | Four minutes
  The Two/2 Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity, particularly for those who cannot manage the longer Six Minute Walk Test (6MWT) or 12 Minute Walk Test.
Pulmonary Function Test | Ten minutes
  Pulmonary function tests (PFTs) allow health proffessionals to evaluate the respiratory function of their patients in many clinical situations and when there are risk factors for lung disease, occupational exposures, and pulmonary toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu Şehir Hastanesi, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared with other researchers.

REFERENCES:
- [Background] Martin-Sanchez C, Calvo-Arenillas JI, Barbero-Iglesias FJ, Fonseca E, Sanchez-Santos JM, Martin-Nogueras AM. Effects of 12-week inspiratory muscle training with low resistance in patients with multiple sclerosis: A non-randomised, double-blind, controlled trial. Mult Scler Relat Disord. 2020 Nov;46:102574. doi: 10.1016/j.msard.2020.102574. Epub 2020 Oct 8. PMID 33296972
- [Background] Huang MH, Fry D, Doyle L, Burnham A, Houston N, Shea K, Smith H, Wiske L, Goode J, Khitrik E, Kolanda M. Effects of inspiratory muscle training in advanced multiple sclerosis. Mult Scler Relat Disord. 2020 Jan;37:101492. doi: 10.1016/j.msard.2019.101492. Epub 2019 Nov 1. PMID 31707233
- [Background] Inzelberg R, Peleg N, Nisipeanu P, Magadle R, Carasso RL, Weiner P. Inspiratory muscle training and the perception of dyspnea in Parkinson's disease. Can J Neurol Sci. 2005 May;32(2):213-7. doi: 10.1017/s0317167100003991. PMID 16018157
- [Derived] Duman Ozkan T, Oguz S, Unal E, Emir C, Polat MG. Effects of inspiratory muscle training on balance, trunk control, fear of falling, respiratory function, and quality of life in people with multiple sclerosis: a randomized controlled trial. Mult Scler Relat Disord. 2025 Nov;103:106699. doi: 10.1016/j.msard.2025.106699. Epub 2025 Aug 18. PMID 40848620